CLINICAL TRIAL: NCT06371001
Title: Prevalance Of Helicobacter Pylori Infection In Chonic Kidney Diseased Patient Admitted To Luxor Medical
Brief Title: Prevalance Of Helicobacter Pylori Infection In Chonic Kidney Diseased Patient Admitted To Luxor Medical Complex
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gehad Abdel Shafy Ahmed Abdel kader, Prevalance Of Helicobacter Pylori Infection In Chonic Kidney Diseased Patient, Assiut University
Other Study IDs: Helicobacter Pyloi and CKD
Record Dates: First submitted 2024-04-13; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- prevalence of helicobacter pylori in chronic kidney diseased patient: prevalence of helicobacter pylori in chronic kidney diseased patient
  Interventions: Other: disease
- prevalence of helicobacter pylori in non chronic kidney diseased patient: prevalence of helicobacter pylori in non chronic kidney diseased patient
  Interventions: Other: disease

INTERVENTIONS:
Other: disease — Helicobacter Pylori Infection In Chonic Kidney Diseased Patien

SUMMARY:
Detect prevalence of Helicobacter pylori infection in chronic kidney diseased patient admitted to Luxor medical complex and possible role of Helicobacter pylori in pathogenesis of chronic kidney diseased patient of unknown etiology

DETAILED DESCRIPTION:
Helicobacter Pylori bacteria is the main pathogenic organism that settles on the gastric mucosa of more than half the human population around the world, with more prominence in the developing countries. H. Pylori had been found to be the main factor in acute and chronic gastritis, peptic ulcer diseases, and in most cases gastric malignancy. Beside to some extra gastro-intestinal diseases. Such as cardiac, pulmonary, renal and hematological diseases.

Another study showed a significant higher proteinuria in H. Pylori infected patients compared to non-infected individuals. Helicobacter pylori is a gram-negative bacterium infecting both children and adults. It is the most common human chronic infection, causing gastrointestinal diseases such as gastric malignancies, gastritis, and ulcerative diseases. H. pylori can also be involved in other non gastrointestinal infections such as diabetes and metabolic syndrome, heart disease, hematologic disorders, cancer, and chronic kidney disease (CKD) as well as chronic renal failure (CRF).

Some chronic renal failure patients who have received hemodialysis for long periods complained of gastrointestinal troubles. It has been postulated that high urea concentration makes the gastric mucosa of these patients more susceptible to H. pylori colonization. Previous observations in different countries reported the prevalence of H. pylori infection among patients with CRF ranging between 20 and 60%, and H. pylori infection can contribute to progressive renal dysfunction resulting in CKD development. In patients without established gastric dysfunction, the presence of H pylori infection was associated with increased risk for Chronic kidney dusease however, patients with both atrophic gastritis (AG) and Helcobacter pylori infection appeared to be at decreased risk for Chronic kidney disease compared with control participants.

For the H. pylori-positive patients with peptic ulcer, H. pylori infection may be a risk factor resulting in kidney damage and H. pylori eradication probably benefits to kidney damage relief and chronic kidney disease prevention.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged >18 years old with chronic kidney disease of different etiology based on clinical examination, laboratory investigations and imaging

Exclusion Criteria:

1. Patients aged ≤18 years old.
2. Overloaded patients
3. patient with acute kidney injury
4. Patients with other GIT disease
5. pregnant female
6. patient taking aspirin, NSAID, steroid or antibiotic
7. Presence of malignancy

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Prevalance Of Helicobacter Pylori Infection In Chonic Kidney Diseased Patient Admitted To Luxor Medical complex hospital
Sampling Method: Non-Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori infection and Chronic kidney diseased patient | 1 year
  Detect prevalence of H pylori infection in chronic kidney diseased patient admitted to Luxor medical complex hospital

SECONDARY OUTCOMES:
possible role of H pylori in pathogenesis of chronic kidney diseased patient of unkown etiology | 1 year
  possible role of H pylori in pathogenesis of chronic kidney diseased patient of unkown etiology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shin SP, Bang CS, Lee JJ, Baik GH. Helicobacter pylori Infection in Patients with Chronic Kidney Disease: A Systematic Review and Meta-Analysis. Gut Liver. 2019 Nov 15;13(6):628-641. doi: 10.5009/gnl18517. PMID 30970438
- [Background] Zizzi CF, Pellicano R, Biancone L. The relationship between Helicobacter pylori and chronic kidney disease: update 2020. Minerva Gastroenterol Dietol. 2020 Dec;66(4):343-349. doi: 10.23736/S1121-421X.20.02729-4. Epub 2020 Jul 3. PMID 32623870
- [Background] Hata K, Koyama T, Ozaki E, Kuriyama N, Mizuno S, Matsui D, Watanabe I, Uehara R, Watanabe Y. Assessing the Relationship between Helicobacter pylori and Chronic Kidney Disease. Healthcare (Basel). 2021 Feb 3;9(2):162. doi: 10.3390/healthcare9020162. PMID 33546229
- [Background] Lin SY, Lin CL, Liu JH, Yang YF, Huang CC, Kao CH. Association between Helicobacter pylori infection and the subsequent risk of end-stage renal disease: a nationwide population-based cohort study. Int J Clin Pract. 2015 May;69(5):604-10. doi: 10.1111/ijcp.12602. Epub 2015 Jan 21. PMID 25644865